CLINICAL TRIAL: NCT00743613
Title: Predicting Peripheral Arterial Disease in Men With Erectile Dysfunction
Acronym: PREPARED
Status: Completed | Type: Observational
Sponsor: Bruton Avenue Family Practice (Other)
Collaborators: Pfizer (Industry)
Responsible Party: James Travers Edwards, Jr., MD Principal investigator, Bruton Avenue Family Practice
Other Study IDs: PREPARED 001
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Erectile Dysfunction; Peripheral Arterial Disease
Keywords: Erectile Dysfunction; ED; Peripheral Arterial Disease; PAD; Ankle-Brachial Index; ABI
MeSH Terms: conditions — Erectile Dysfunction; Peripheral Arterial Disease | interventions — Menogaril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Sexual Health Inventory for Men (SHIM) — Five question test with maximum score of 25 points administered on the initial visit. Erectile dysfunction is indirectly related to the score.
  Other Names: SHIM; Sexual Health Inventory for Men
Procedure: Ankle-Brachial Index (ABI) — Measure Ankle-Brachial Index with a hand held doppler and sphygmomanometer to determine the ABI.
  Other Names: Multi Dopplex II 8-mHz

SUMMARY:
Erectile dysfunction is a common complaint and is found frequently in men with hyperlipidemia, hypertension, diabetes and those who smoke. ED may also be an early warning of peripheral arterial disease. This study is designed to look for a relationship between the degree of ED and the presence of PAD when associated with co-morbid conditions.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is a common complaint in the primary care office. It is frequently found in men with hyperlipidemia, hypertension, or diabetes, and may also be an early warning of peripheral arterial disease. We looked for a relationship between the degree of ED and the presence of PAD as measured by the Ankle Brachial Index (ABI) associated with co-morbid conditions. Men over the age of 50 with hyperlipidemia, diabetes, hypertension, or tobacco use were asked to complete a Sexual Health Inventory for Men (SHIM). An ABI was measured using a hand held Doppler. 175 men from two urban and three suburban Family Practices in Tidewater Virginia participated. Outcome measures included SHIM scores, ABI, Systolic Blood Pressure, LDL, Hemoglobin A1C and tobacco use. Moderate or severe erectile dysfunction (SHIM < 11.0) was identified in 44% of participants. More than 12.5% of men with severe ED (SHIM < 7.0) had an ABI positive for PAD at 0.95 or less. The results were adjusted for the presence of hyperlipidemia, hypertension, diabetes and tobacco use. Men with hypertension did not demonstrate a significant increase in the frequency of PAD compared to diabetics or smokers. Neither race nor age was found to increase the prevalence of ED. The complaint of erectile dysfunction in men over age 50 should prompt a physician to consider peripheral arterial disease. A simple self-administered SHIM test should help identify men at risk for PAD and suggest further evaluation if the score is 7.0 or less.

ELIGIBILITY:
Inclusion Criteria:

* Men 50 years old or older
* Must have a history of diabetes, hypertension, hyperlipidemia and/or a history of tobacco use

Exclusion Criteria:

* Men younger than 50 years of age
* No co-morbid condition such as diabetes, hypertension, hyperlipidemia and/or tobacco use.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men 50 years old or older with either diabetes, hypertension, hyperlipidemia and/or a history of tobacco use.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2005-02; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Sexual Health Inventory for Men (SHIM) | initial visit

SECONDARY OUTCOMES:
Ankle-Brachial Index (ABI) | Initial Visit

CONTACTS AND LOCATIONS:
Overall Officials: James T Edwards, Jr, MS, MD, Principal Investigator — Bruton Avenue Family Practice
Locations (5):
- United States (5):
  - UMass, Fitchburg Family Medicine Center, Fitchburg, Massachusetts
  - Mercury West Family Practice, Hampton, Virginia
  - Bruton Avenue Family Practice, Newport News, Virginia
  - Hilton Family Practice, Newport News, Virginia
  - Williamsburg Medical Arts-Family Medicine, Williamsburg, Virginia

REFERENCES:
- [Result] Grover SA, Lowensteyn I, Kaouache M, Marchand S, Coupal L, DeCarolis E, Zoccoli J, Defoy I. The prevalence of erectile dysfunction in the primary care setting: importance of risk factors for diabetes and vascular disease. Arch Intern Med. 2006 Jan 23;166(2):213-9. doi: 10.1001/archinte.166.2.213. PMID 16432091
- [Result] Gazzaruso C, Giordanetti S, De Amici E, Bertone G, Falcone C, Geroldi D, Fratino P, Solerte SB, Garzaniti A. Relationship between erectile dysfunction and silent myocardial ischemia in apparently uncomplicated type 2 diabetic patients. Circulation. 2004 Jul 6;110(1):22-6. doi: 10.1161/01.CIR.0000133278.81226.C9. Epub 2004 Jun 21. PMID 15210604
- [Result] Lue TF. Erectile dysfunction. N Engl J Med. 2000 Jun 15;342(24):1802-13. doi: 10.1056/NEJM200006153422407. No abstract available. PMID 10853004
- [Result] Solomon H, Man JW, Jackson G. Erectile dysfunction and the cardiovascular patient: endothelial dysfunction is the common denominator. Heart. 2003 Mar;89(3):251-3. doi: 10.1136/heart.89.3.251. PMID 12591819
- [Result] Jackson G. Endothelial function and dysfunction. Int J Clin Pract. 2004 May;58(5):431. doi: 10.1111/j.1368-5031.2004.00255.x. No abstract available. PMID 15206495
- [Result] Deedwania PC. Endothelium: a new target for cardiovascular therapeutics. J Am Coll Cardiol. 2000 Jan;35(1):67-70. doi: 10.1016/s0735-1097(99)00536-7. No abstract available. PMID 10636261
- [Result] Hurairah H, Ferro A. The role of the endothelium in the control of vascular function. Int J Clin Pract. 2004 Feb;58(2):173-83. doi: 10.1111/j.1368-5031.2004.0103.x. No abstract available. PMID 15055866
- [Result] Kloner RA. Erectile dysfunction in the cardiac patient. Curr Urol Rep. 2003 Dec;4(6):466-71. doi: 10.1007/s11934-003-0028-9. PMID 14622500
- [Result] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Result] Cappelleri JC, Rosen RC. The Sexual Health Inventory for Men (SHIM): a 5-year review of research and clinical experience. Int J Impot Res. 2005 Jul-Aug;17(4):307-19. doi: 10.1038/sj.ijir.3901327. PMID 15875061
- [Result] Sutton-Tyrrell K, Rihal C, Sellers MA, Burek K, Trudel J, Roubin G, Brooks MM, Grogan M, Sopko G, Keller N, Jandova R. Long-term prognostic value of clinically evident noncoronary vascular disease in patients undergoing coronary revascularization in the Bypass Angioplasty Revascularization Investigation (BARI). Am J Cardiol. 1998 Feb 15;81(4):375-81. doi: 10.1016/s0002-9149(97)00934-x. PMID 9485122
- [Result] Carman TL, Fernandez BB Jr. A primary care approach to the patient with claudication. Am Fam Physician. 2000 Feb 15;61(4):1027-32, 1034. PMID 10706155
- [Result] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Result] Champion H. Erectile Dysfunction and Cardiovascular Disease: Carrots, Sticks, and Better Men's Health. Adv Stud Med. 6(4):163-170, 2006
- [Result] Vinick A, Richardson D. Erectile Dysfunction in Diabetes. Diabetic Reviews 6:16-33, 1998.
- [Result] Fedele D, Bortolotti A, Coscelli C, Santeusanio F, Chatenoud L, Colli E, Lavezzari M, Landoni M, Parazzini F. Erectile dysfunction in type 1 and type 2 diabetics in Italy. On behalf of Gruppo Italiano Studio Deficit Erettile nei Diabetici. Int J Epidemiol. 2000 Jun;29(3):524-31. PMID 10869326
- [Result] Brunton S: Raising the Profile of Peripheral Arterial Disease. AANP 18th Annual National Conference, July 1, 2003, Anaheim, CA.